CLINICAL TRIAL: NCT00974415
Title: A Pilot Study of the Carbon Dioxide Treatment for Fat Reduction
Brief Title: Study of the Carbon Dioxide Treatment for Fat Reduction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STU11387
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Overweight
Keywords: BMI classification-overweight
MeSH Terms: conditions — Overweight | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment (Experimental): CO2 treatment
  Interventions: Procedure: CO2
- sham (Sham Comparator): sham treatment
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: CO2 — CO2 treatment delivered to randomized flank at each study visit
  Arms: treatment
Procedure: Sham — Sham treatment to other flank at each study visit
  Arms: sham

SUMMARY:
The primary objective of this study is to demonstrate the efficacy and safety of the carbon dioxide for subcutaneous fat reduction.

ELIGIBILITY:
Inclusion criteria:

* Male or female subject ages ≥ 18 years old
* Body mass index (BMI) between 18.5-24.99. (BMI is defined as weight in pounds multiplied by 703 divided by the square of the height in inches).

Subject in good health

* Willing and able to abstain from partaking in any treatment other than the study procedure (existing or new) to promote body contouring and/or weight loss during the course of study participation.
* Subject agrees to maintain their weight (i.e. within 5 pounds) by not making any changes to diet or lifestyle during the study.
* The subject has the willingness and the ability to understand and provide informed consent for the use of their tissue and communicate with the investigator

Exclusion criteria:

* Pregnant or lactating or intends to become pregnant in the next 9 months.
* Unable to understand the protocol or to give informed consent
* Any previous and/or pending procedures at the treatment area or that may likely affect the treatment area
* Pending and/or anticipated major change in diet or exercise pattern in the six weeks following the last treatment or who has taken diet pills within the last 6 months.
* History of asthma or chronic obstructive pulmonary diseases
* Active skin disease or skin infection in the treatment area
* Bleeding tendency or coagulopathy
* Subject who are allergic to lidocaine
* Any other condition that would, in the professional opinion of the investigator, potentially affect response or participation in the clinical study, or would pose as an unacceptable risk to the subject

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2010-01; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of flank circumference | 6 months

SECONDARY OUTCOMES:
10-point pain visual analog scale | 4 weeks
Any adverse events | 6 months
Patient satisfaction, determined by using patient satisfaction questionnaires. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States